CLINICAL TRIAL: NCT06543433
Title: Skincubator (Model 2), a Novel Incubator for Skin to Skin Contact Feasibility Study, in Monash and Riverside
Brief Title: Skincubator, a Novel Incubator for Skin to Skin Contact Feasibility Study
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Itamar Nitzan (Other)
Collaborators: Monash University (Other); Monash Health (Other); Riverside University Health System Medical Center (Other)
Responsible Party: Sponsor-Investigator, Itamar Nitzan, Dr, Shaare Zedek Medical Center
Organization: Shaare Zedek Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: V1 15.5.2024
Record Dates: First submitted 2024-08-03; First posted 2024-08-09 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Preterm; Preterm Birth
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Intervention Model Description: The intervention will be given to all participants and the investigators will test how many hours of SSC per day the parents can achieve.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Skincubator (Experimental): This is the only arm. All babies in trial will receive the intervention.
  Interventions: Device: Skincubator 2

INTERVENTIONS:
Device: Skincubator 2 — The Skincubator is a small incubator designed to attach to the caregiver's torso without any barrier between the parent's chest and the baby. It creates an environment with the advantages of a standard neonatal incubator, while enabling Skin to Skin contact for extended periods from birth. It has multiple access points, to allow for common nursing procedures. It is anchored safely to the parent's body and secures ventilator and IV tubing. It also includes side ports for the parents to insert their hands to touch their baby.
  The investigators will offer the parents in the intervention group the opportunity to perform Skincubator care for as long as they want to each day during the week after enrolment. The investigators will provide the parents with the aids to accomplish this goal: the Skincubator system with a convenient environment, the option for Skincubator surrogates and, where possible, the option for one of the parents to sleep with the baby safely secured in the Skincubator.

SUMMARY:
The goal of this clinical trial is to test the feasibility of using the Skincubator, a wearable incubator for skin to skin contact of preterm babies and their parents. It will also learn about the safety of skincubator. The main questions it aims to answer are:

* Can the Skincubator keep a stable temperature for the smallest babies and the first days after birth?
* How many hours will the parents (and other family members) will succeed to perform skin to skin every day?

Participants will:

Be offered the opportunity to perform Skincubator care for as long as they want to each day during the week after enrolment.

DETAILED DESCRIPTION:
Study design: This is a non-randomized feasibility trial with no control group in which the investigators will offer parents the option to perform Skincubator care - being cared for in SSC inside the Skincubator, which is placed on the mother and/or another caregiver. Skincubator care will be provided from birth if the caring team and the parents feel it is appropriate. The option for Skincubator care will be provided for as long as the parents, surrogates, and staff feel comfortable with a goal of possible achievement of the WHO target of 8 hours per day. Each infant will participate in the study for one week from enrollment (If parents desire, they will be able to continue using the Skincubator beyond 1 week as long as NICU staff feel that it is helpful for the baby).

Implementation phase: Prior to beginning the study, each center will provide care in the Skincubator for five noninvasively ventilated preterm babies. After gaining experience in treating a preterm baby in the Skincubator and performing manikin simulations of Skincubator care for invasively ventilated babies, the NICU team in each center will be able to decide whether to include intubated babies in the trial.

Population: up to 25 preterm neonates in each site, born at GA of 24.0-32.6 with birth weight of <1.5 kg.

First 3 babies will be of GA of 26-32.6 and on noninvasive respiratory support. Those babies will be considered a learning phase for the team, and may be analyzed separately. After completing the learning phase the study will proceed with 4 groups:

1. Up to 7 more babies of GA of 26-32.6 and on noninvasive respiratory support.
2. 5 Intubated babies with GA of 26-32.6. The investigators will start enrolling babies from this group only after the team treated at least 5 babies from group 1 (including the learning phase) and feels ready to move on to intubated babies.
3. 5 babies GA 24.0-25.6 on noninvasive respiratory support. The investigators will start enrolling babies from this group only after the team treated at least 5 babies from group 1 (including the learning phase) and feels ready to move on to this age group.
4. 5 intubated babies with GA of 24.0-25.6. The investigators will start enrolling babies from this group only after the team treated at least 3 babies from group 2 and 3 babies from group 3, and only if the team feels ready to move on to this group also.

First five babies will be treated in the Skincubator only from NICU admission. After gaining experience with the first 5 babies the team may decide to start Skincubator care in birth suite (ideally on the mother, potentially on the father if the mother prefers or is feeling unwell) or in cesarean section theater (on the father).

ELIGIBILITY:
Inclusion Criteria:

* Preterm neonates with birth weight of <1.5 kg
* Requiring respiratory support
* Cared for in an incubator with at least 60% humidity.

Exclusion Criteria:

* Critical congenital heart disease
* Suspected genetic syndrome
* Hemodynamic instability
* Having a chest tube,
* Significant congenital anomalies,
* Need for surgery
* If the attending neonatologist decides that the Skincubator is not safe for a specific baby.
* Neonates whose mothers have a significant mental disorder that is not adequately controlled
* Neonates of parents unable to perform extended SSC for any reason will be excluded as well.

Ages: 0 Days to 14 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2024-08-31 (Estimated); Primary Completion 2026-09-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
hours of SSC per day | In the first week from study commencement (study commencement will be defined as birth or receiving consent, whichever occurs later).
  primary neonatal outcome will be hours of SSC per day
Parental Stress Scale (PSS) NICU | 4 to 7 days after birth.
  Parental Stress Scale (PSS) NICU performed by the mother. Minimum and maximum values for PSS NICU are 0 and 72, higher scoring indicates higher parental stress.

SECONDARY OUTCOMES:
Time outside of temperature range 36.5-37.5 | In the first week from study commencement (study commencement will be defined as birth or receiving consent, whichever occurs later).
  Time outside of temperature range 36.5-37.5 measured axillary
time in environmental humidity of less than 60% | In the first week from study commencement (study commencement will be defined as birth or receiving consent, whichever occurs later).
  time in environmental humidity of less than 60% measured by hygrometer and incubator hygrometer

CONTACTS AND LOCATIONS:
Overall Officials: Itamar Nitzan, M.D, Study Director — Shaare Zedek Medical Center
Locations (1):
- Monash Children's hospital, Clayton, Victoria, Australia

IPD SHARING:
Plan to Share IPD: Undecided
The investigators will need to discuss with local IRBs